CLINICAL TRIAL: NCT05338567
Title: Digital Three-dimensional Reconstruction for Predicting Small Bowel Length in Bariatric Surgery
Brief Title: Digital 3D Reconstruction Predicts Small Bowel Length
Acronym: DTDRPSBL-BS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, fan li, DapingH, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: 3DRABL-BS
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Small Intestine Length Measurement
Keywords: bariatric surgery; Roux-en-y gastric bypass; Type 2 diabetes mellitus; Three-Dimensional reconstruction
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open/laparoscopic surgery: Small bowel length measurement by laparoscopy or laparotomy
- 3D reconstruction: Small bowel length measurement by 3D digital model
  Interventions: Diagnostic Test: Small intestine length measurement method

INTERVENTIONS:
Diagnostic Test: Small intestine length measurement method — Accuracy of digital 3D reconstruction for predicting small bowel length
  Groups: 3D reconstruction

SUMMARY:
The prevalence of type 2 diabetes mellitus (T2DM) has been increasing annually worldwide, and the prevalence of diabetes has reached 11.6% in China. Laparoscopic Roux-en-Y gastric bypass (RYGB) is still widely accepted as a valid surgery in the treatment of obesity and T2DM. But still, there is no consensus on the ideal of the gastric bypass limb lengths. Reported lengths of biliopancreatic limb (BPL) and alimentary limb (AL) varied widely from 10-250 to 35-250 cm, and anatomical data show that the length of small intestine varies greatly among adults. Choosing the same small bowel bypass length for different individuals obviously cannot achieve the expected weight loss effect, and individuals with too short small intestine can cause severe malnutrition complications and even life-threatening conditions. Therefore, measurement of small bowel length is one of the prerequisites for performing precise RYGB. Intraoperative measurement of small bowel length can increase the operative time and the risk of surgical complications such as intestinal perforation. So, predicting the total length of the small intestine is very important for accurately performing bariatric surgery and avoiding the risk of surgical complications. In this study, we propose to perform 3D segmentation and reconstruction of the small intestine by acquiring abdominal CT data through digital technology, and predict the small intestine length by 3D digital measurement of the small intestine, and verify the digital measurement data by performing digital measurement data. Establish a small bowel length prediction model for bariatric surgery to develop a more accurate and personalized gastric bypass surgery plan for patients to obtain weight loss and glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for surgical treatment of T2DM were selected based on the Chinese Guidelines for the Surgical Treatment of Obesity and Type 2 Diabetes (2019 )

Exclusion Criteria:

* Adhesions, peritonitis, and patients who have had bowel resection (small intestine, colon or rectum) that hinder the measurement of the entire intestinal length
* Non-weight loss surgery patients whose incision is less than 6 cm are not suitable for measuring the length of the small intestine.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent bariatric surgery in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2023-10-02 (Estimated); Study Completion 2023-10-02 (Estimated)

PRIMARY OUTCOMES:
Validation of the accuracy of the predicted length of the small intestine | 2 years
  The accuracy of the 3D reconstruction method was judged by comparing the length of the small intestine measured by the open/laparoscopic surgery with the length of the small intestine calculated by the preoperative CT 3D reconstruction.

SECONDARY OUTCOMES:
Building prediction formulas through machine deep learning | 2 years
  Through robotic deep learning, the small intestine is automatically segmented, and the small intestine is reconstructed in three dimensions to calculate the length of the small intestine.

CONTACTS AND LOCATIONS:
Overall Officials: fan Li, PhD, Study Director — Army medical universtiy daping hospital
Locations (1):
- Daping hospital, Chongqing, China

IPD SHARING:
Plan to Share IPD: No